CLINICAL TRIAL: NCT04515472
Title: Effect of Gender Affirming Hormone Therapy on Glucose Metabolism
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: VA policy released 3/17/25 to phase out treatment for gender dysphoria
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Foundation for Advancing Veterans' Health Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20190415H
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Transgender Persons
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Intervention Model Description: MTF and FTM non-diabetic transsexuals will be compared to healthy female and male subjects respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteer Male (Active Comparator): Healthy male currently on no testosterone treatment
  Interventions: Drug: Botnia Clamp
- Healthy Volunteer Female (Active Comparator): Healthy female currently on no estrogen treatment
  Interventions: Drug: Botnia Clamp
- MTF group (Active Comparator): MTF transgender currently on estrogen treatment
  Interventions: Drug: Botnia Clamp; Other: Withdrawal of Gender Affirming Hormone Therapy (GAHT)
- FTM group (Active Comparator): FTM transgender group currently on testosterone treatment
  Interventions: Drug: Botnia Clamp; Other: Withdrawal of Gender Affirming Hormone Therapy (GAHT)

INTERVENTIONS:
Drug: Botnia Clamp — This clamp technique is designed to obtain independent measures of insulin secretion and insulin sensitivity during the same test. In brief, 0.3g/kg body wt of a 20% glucose solution is given at time 0. Blood samples for the measurement of plasma glucose and serum insulin are obtained at -10, 0, 2, 4, 6, 8, 10, 20, 30, 40, 50, 60, 120, and 180 min.
  Other Names: Glucose solution and insulin
Other: Withdrawal of Gender Affirming Hormone Therapy (GAHT) — GAHT, either estrogen or testosterone therapy will be withdrawn after the Botnia Clamp.
  Arms: FTM group; MTF group

SUMMARY:
The study will test:

1. whether estrogen treatment in transwomen is associated with improved insulin sensitivity and beta cell function
2. whether testosterone treatment in transmen is associated with worsening insulin sensitivity and beta cell function
3. whether estrogen therapy leads to enhanced immune response in older transwormen

DETAILED DESCRIPTION:
All subjects will participate in a 2-hour oral glucose tolerance test (OGTT) and DXA scan for estimation of lean body mass. Only the transgender subjects will have a repeat OGTT two weeks after discontinuation of Gender Affirming Hormone Therapy (GAHT).

Beta cell function will be correlated with the Estrogen/Testosterone ratio to evaluate the relationship between sex hormones and beta cell function. Plasma Glucagon-like peptide 1 (GLP-1) response during the OGTT will be measured to evaluate if estrogen treatment modulates insulin secretion by increasing GLP-1 secretion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: healthy male or female
* MTF transgender
* FTM transgender
* Non-diabetic (A1c<6.5%), fasting glucose <126mg/dl and OGTT after 2 hr <200mg/dl)
* Stable hormone treatment (estrogen or testosterone) for at least 6 months

Exclusion Criteria:

* History of or newly diagnosed diabetes mellitus
* For healthy volunteers, not current treatment with estrogen or testosterone
* For FTM transgender, no recent cardiovascular event: acute coronary syndrome (ACS), stroke (CVA)
* For MTF and FTM transgender, less than 6 months of stable hormone treatment
* Anemia with hemoglobin (Hb) <11.0 hematocrit (Hto) < 34 and Glomerular Filtration rate (GFR) <30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Effects of Chronic estrogen therapy on insulin secretion | Baseline to 180 minutes
  Change in GLP-1 in response to glucose
Effects of Chronic estrogen therapy on insulin sensitivity | Baseline to 6 months
  Change in beta cell function
Effects of Chronic testosterone therapy on insulin secretion | Baseline to 180 minutes
  Change in GLP-1 in response to glucose
Effects of Chronic testosterone therapy on insulin sensitivity | Baseline to 6 months
  Change in beta cell function

SECONDARY OUTCOMES:
Immune response change | Baseline to 6 months
  Withhold GAHT for 2 weeks after Botnia Clamp

CONTACTS AND LOCATIONS:
Overall Officials: Devjit Tripathy, MD, Principal Investigator — University of Texas Health San Antonio
Locations (1):
- Bartter Clinical Research Unit, Audie L. Murphy VA Hospital, sTXVHCS, San Antonio, Texas, United States